CLINICAL TRIAL: NCT05416255
Title: Measuring Synovial Fluid Components
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dharma Bioscience (Other)
Responsible Party: Principal Investigator, Gastón Andres Topol, Treating physician and primary investigator, Dharma Bioscience
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFComponents#1
Record Dates: First submitted 2022-06-05; First posted 2022-06-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Consecutive patients treated for knee osteoathritis with dextrose injection, hemaopoietic stem cell injection, PRP injection, or no injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dextrose injection (Active Comparator): Injection of 10 ml of 12.5% dextrose
  Interventions: Diagnostic Test: Measuring synovial fluid components
- Hematopoietic stem cells (Active Comparator): Injection of 10 ml of of 7.5 ml hematopoietic stem cells, 2 ml of 25% dextrose (5% diluted), 0.5 ml of 1% lidocaine (0.05% diluted),and 0.25 ml dexamethasone (1.5 mg)
  Interventions: Diagnostic Test: Measuring synovial fluid components
- Platelet Rich Plasma injection (Active Comparator): Injection of 10 ml of leukocyte rich platelet rich plasma
  Interventions: Diagnostic Test: Measuring synovial fluid components
- No injection (Active Comparator): Aspiration of synovial fluid may be an active comparator.
  Interventions: Diagnostic Test: Measuring synovial fluid components

INTERVENTIONS:
Diagnostic Test: Measuring synovial fluid components — Using speialized techniques to measure S.F. components

SUMMARY:
Participants with grade 3 and 4 knee osteoarthritis will recieve aspiration of synoivial fluid, and then receive either dextrose, hemaotopoietic stem cell, or platelet rich plasma, or no injection. The synovial fluid will be analyzed for changes in components.

DETAILED DESCRIPTION:
80 participants with grade 3 and 4 symptomatic knee osteoarthritis, with a visable effusion, will receive aspiration of 3 ml of synovial fluid from the suprapatellar pouch, followed by either injection with 10 mL of 12.5% dextrose, 10 cc hematopoietic stem cells, 10cc PRP, or no injection into the suprapatellar pouch. They will then receive aspiration of 3 ml of synovial fluid at 2 days and either 7 days (for dextrose injected or no injection) or 14 days (stem cell and PRP injected) days post injection. These synovial samples will be analyzed for a change in components.

ELIGIBILITY:
Inclusion Criteria:≥ 6 months of knee pain with walking

* ≥ 6/10 on a 0-10 point numerical rating scale
* High grade medial compartment cartilage loss ( Kellgren-Lawrence grade 3 or 4) on plain weight bearing X-ray
* Exposed subchondral bone at 110 degrees of flexion by ultrasound examination
* Easily visible suprapatellar pouch with quads conttraction.

Exclusion Criteria

* Current intake of NSAIDs or steroids
* Current anticoagulation therapy
* Inflammatory or post-infectious knee arthritis
* Systemic inflammatory conditions
* Knee flexion less than 100 degrees
* Knee extension less than 165 degrees
* Valgus or varus more than 15 degrees
* Any knee injection in the precedign 3 months
* BMI more than 50 kg/ meter squared
* Gross synovial folds on ultrasound.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine and unspecified component levels in synovial fluid | Day 0 to Day 14
  Change in level of unspecified synovial fluid components from Day 0 to 7 or Day 0 to 14, depending on group

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) (0-100 scale) Higher scores are a worse outcome. | Day 0 to Day 14
  Change in WOMAC score from Day 0 to Day 14

OTHER OUTCOMES:
0-10 Numerical Rating Scale for pain (NRS) (11 point scale. Higher values are a worse outcome) | Day to Day 14
  Change in NRS pain score from Day 0 to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Dharma Centro de Medicina Regenerativa, Rosario, Santa Fe Province, Argentina